CLINICAL TRIAL: NCT04525924
Title: Feasibility Study of Adjunctive Bright Light Therapy (BLT) for Amelioration of Fatigue in Chinese Cancer Patients Admitted to a Palliative Care Unit
Brief Title: Feasibility of Adjunctive BLT for Amelioration of Fatigue in Chinese Cancer Patients Admitted to a Palliative Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Tang Heng Joshua, Deparment of Medicine & Geriatrics, Resident, Principal Investigator, Hospital Authority, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FatigueBLT
Record Dates: First submitted 2020-07-28; First posted 2020-08-25 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Fatigue; Cancer
Keywords: fatigue; cancer; palliative care; BLT; bright light therapy; feasibility
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bright light therapy (Experimental): Bright light therapy (BLT) will be given via a lightbox device in the morning for 30 minutes after waking up. Duration of therapy will be 7 consecutive days.
  Interventions: Device: bright light therapy

INTERVENTIONS:
Device: bright light therapy — please see arm description

SUMMARY:
Fatigue is the most common symptom in palliative care patients who have advanced cancer. Fatigue is also one of the most underreported hence under-treated symptoms. Patients may perceive it as a condition to be endured, whereas healthcare workers find it very challenging to assess and treat due to its subjective nature and multi-dimensional causes.

However, evidence-based practice to tackle this distressing problem is still inadequate, and that a one-size fit all approach is unrealistic. Various pharmacological options have been examined, but due to limited evidence, no specific drug could be recommended.

Latest development in management of fatigue includes non-pharmacological approach. Bright Light Treatment (BLT) has also evolved as a favourable treatment for cancer-related fatigue. BLT is the prescription of artificial bright light over a designated period of time. Recent clinical evidence showed that BLT reduced symptom of fatigue in patients undergoing active chemotherapy and cancer survivours.

There is however no data on bright light therapy used in in-patient palliative care settings.

A single group, prospective interventional study will be conducted in in-patient palliative care unit of Shatin Hospital (N = 42). The aim is to assess the feasibility and impact of BLT as an in-patient intervention in a cohort of local Chinese palliative care in-patients diagnosed with incurable cancer with documented symptom of fatigue, and to ascertain the changes of fatigue, mood, sleep and quality of life after 1-week exposure of BLT.

DETAILED DESCRIPTION:
Fatigue is the most common symptom in palliative care patients who have advanced cancer, ranging from 59% to 77% depends on the assessment method (1). There is limited local data on the prevalence of fatigue in cancer patients. A cross-sectional study by Dr KY Lam in 2009 (unpublished data) found 53% of 55 patients receiving palliative care suffered from severe fatigue. A cross-sectional symptom screening of all the patients in the palliative care ward in Shatin Hospital showed 22 out of 55 (40%) patients reported fatigue (unpublished data).

The fatigue experienced by cancer patients is multi-dimensional. The feeling may be a physical sensation (weakness, tiredness, exhaustion, unable to perform tasks), an affective sensation (low mood, lack of motivation), or a cognitive sensation (lack of concentration, difficulty thinking clearly). This phenomenon is also subject to cultural interpretation therefore there is a need to understand each subject's perception and experience of fatigue within his or her own cultural context (2, 3).

Fatigue is also one of the most under-reported hence under-treated symptoms. Patients may perceive it as a condition to be endured, whereas healthcare workers find it very challenging to assess and treat due to its subjective nature and multidimensional causes. The impairment in self-care capabilities and daily functioning lead to negative effects on desire to continue treatment thus affecting the functional recovery even in patients with a more stable disease status (3-5). The quality of life (QOL) of patients, which is our focus in palliative care service, is heavily reduced (6).

However, evidence-based practice to tackle this distressing problem is still inadequate, and that a one-size fit all approach is unrealistic (7). Various pharmacological options have been examined, but due to limited evidence, no specific drug could be recommended for the treatment of fatigue in palliative care patients in the latest Cochrane review in 2015 (8).

Latest development in management of fatigue includes non-pharmacological approach. Effect size in reducing fatigue in various treatments were summarised in a report by Bower (9). Exercise was more effective than control in reducing fatigue with a mean effect size of -0.27. Psychosocial intervention trials that included fatigue as a primary or secondary outcome have shown reductions in fatigue relative to control, with effective sizes ranging from -0.10 to -0.31. Psychostimulant trials, most of which were conducted among patients with advanced disease and used methylphenidate, suggested that psychostimulants were more effective than placebo in improving fatigue with an effect size of -0.28. Of note, two studies with larger sample size showed no benefit for methylphenidate vs. placebo for improving fatigue (10, 11). The application of non-pharmacological approach in our local patients was even more limited. A pilot study of 26 patients receiving palliative care in Shatin Hospital showed a mean change score of 0.5 (1.862) of improvement in Brief Fatigue Inventory (BFI) Q3 after two weeks of in-patient multidisciplinary care (unpublished data). The estimated effect size of the pilot study was 0.268 (mean change/SD = 0.5/1.863). Overall, these data suggest that non-pharmacological treatments (e.g. exercise, psychoeducation, support program, cognitive-behavioural therapy) have a mild to moderate effect on improving symptom of fatigue.

Over these few decades, Bright Light Treatment (BLT) has also evolved as a favourable treatment for cancer-related fatigue. BLT is the prescription of artificial bright light over a designated period of time. It was initially developed for the treatment of seasonal affective disorder, and found to be as effective as antidepressants for treatment of depressive symptoms during winter (12). The National Comprehensive Cancer Network (NCCN) guidelines on cancer-related fatigue (13) and a recent review on all treatment options of cancer-related fatigue (14) suggested that BLT is a safe and accessible option.

There are several mechanisms on how light therapy works. Firstly, it works through improving alertness. Healthy subjects who had increasing bright light exposure as compared to dim light would have a rapid effect of decrease in sleepiness and improvement in their performance (15). Secondly, BLT works through improving mood. Efficacy of BLT have been demonstrated in seasonal affective disorder (12), non-seasonal depression (16) and bipolar depression (17). Thirdly, BLT works through regulation of circadian rhythm. Circadian disruptions were demonstrated in 55 community-dwelling cancer patients receiving palliative care (18). Although the cause and effect between exacerbated fatigue and decreased light exposure could not be confirmed, increased fatigue was significantly correlated with decreased light exposure among patients with breast cancer (19). Exposure to bright light in the morning leads to an advance of endogenous circadian rhythms that results in a realignment of these rhythms with the individual's sleep-wake cycle. Therefore, possibly by providing a corrective phase advance with morning BLT, rhythm dysregulation could be corrected resulting in a reduction of fatigue symptom.

Two trials investigated the impact of light therapy on fatigue and QOL in the same group of 39 women with breast cancer undergoing active chemotherapy (20, 21). Results suggest that morning bright light treatment helped prevent the typical worsening of fatigue and quality of life during chemotherapy treatment. Although the light treatment did not improve overall fatigue in this sample, the lack of deterioration in total fatigue during a period where symptoms typically worsen was encouraging. Another study sought to determine the effect of bright light treatment on cancer-related fatigue among 36 post-treatment survivors (22). At the end of the treatment period, patients who had received bright white light therapy were no longer clinically fatigued, whereas 55% of the patients in the active control condition continued to report clinical fatigue. The effects of the bright white light treatment were maintained 3-weeks post-intervention.

A more recent study again focused on cancer survivors (23, 24). The total fatigue score using the Multidimensional Fatigue Symptom Inventory-Short Form showed an effect size of 1.20 in the bright-white-light intervention group and an effect size of 0.93 in the supposing placebo arm dim-red-light group. These were large within group effect size. This study employed BLT as an adjunctive therapy and the participants were not excluded for using their usual medications (including psychotropic medications). A randomised controlled trial in 2007 reported that selective serotonin reuptake inhibitor (SSRI) do not appear to have beneficial effects on cancer-related fatigue, supporting the distinction between fatigue and depression in cancer patients and suggesting that fatigue is not solely a symptom of depression (25).

Bruera and team tried to introduce BLT to patients with advanced cancer and insomnia in out-patient settings (26). One shortcoming of their study was partly due to a high attrition rate especially in the control arm where dim red light was used as placebo. They suggested future studies to incorporate alternative trial designs to improve the adherence.

There is however no data on bright light therapy used in in-patient palliative care settings. Conducting research on patients receiving palliative care has been particularly challenging (27, 28). Barriers include the difficulty in participation due to limitations of serious illness, complex symptoms and clinical instability, resulting in high attrition and missing data. The MOREcare Statement (29) suggested researchers to use measures which are as short and simple as possible.

Despite these limitations, the present evidence suggests that BLT, a safe and easily delivered treatment, may be a clinically feasible and effective intervention to reduce symptom of fatigue in cancer palliative care patients during hospital stay. This study aims to test the feasibility of administering bright light therapy in cancer palliative care patients for the treatment of fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 years old or above
* Chinese ethnic group
* Diagnosis of incurable cancer
* A score of >=3 in Brief Fatigue Inventory after a period of standard care

Exclusion Criteria:

* Patients who are imminently dying
* Patients who are undergoing chemotherapy or radiotherapy
* Patients who have history of epilepsy, brain tumour, brain metastasis
* Patients who are blind or have retinal disease
* Patents who have photosensitive skin condition
* Patients who have history of bipolar disorder as BLT has been suggested to increase the risk of manic swing in patients with bipolar disorder
* Patients who have their dosage of antidepressants adjusted within 6 weeks
* Patients who have difficulties to communicate effectively
* Patients with impaired mental status precluding the completion of the questionnaire (AMT <5)
* Patients who are unable to give valid consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Rate of declined particilation in the study | At screening stage
  Rate of approached potential subjects who declined participation in the study
Attrition rate | 1 week of the intervention
  Rate of subject drop out (all cause)
Change in brief fatigue inventory | Pre- and post- the 1-week intervention
  Change of scoreing of the brief fatigue inventory (BFI) from baseline to end of treatment. BFI is a 9-item questionnaire measured in 11-point Likert scale. It evaluates the level of present, overall and worst fatigue together with its interference to patients' general activity, mood, walking ability, normal work, relationships with other people and enjoyment of life during the past 24 hours. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index | Pre- and post- the 1-week intervention
  Change in Pittsburgh Sleep Quality Index (PSQI) from baseline to end of treatment. PSQI is a 19-item self-report measure to assess sleep quality. It consists of 7 components measuring duration of sleep, sleep disturbance, sleep latency, day dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and whether a person needs medications in order to sleep. A global score > 5 indicates that a patient reports severe difficulties in at least 2 domains or moderate difficulties in more than 3 areas.
Change in Hospital Anxiety and Depression Scale | Pre- and post- the 1-week intervention
  Change in Hospital Anxiety and Depression Scale (HADS) from baseline to end of treatment. HADS is comprised of 14 questions which assess level of depression and anxiety. Each item is scored from 0-3, thus the patient can score between 0-21 for either anxiety or depression. A literature review identified a cut-off point of 8/21 for anxiety or depression.
Change in McGill Quality of Life Questionnaire - Hong Kong | Pre- and post- the 1-week intervention
  Change in McGill Quality of Life Questionnaire - Hong Kong (MQOL-HK) from baseline to end of treatment. It assesses a patient's QOL in 5 domains (physical, psychological, existential, support and sexual functioning). The physical symptoms subscale allows patients to describe their 3 most disturbing symptoms and rate them. Patients can also rate their perceived QOL as a single item score. Responses are measured in 11-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Joshua Tang, Principal Investigator — Hospital Authority
Locations (1):
- Shatin Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teunissen SC, Wesker W, Kruitwagen C, de Haes HC, Voest EE, de Graeff A. Symptom prevalence in patients with incurable cancer: a systematic review. J Pain Symptom Manage. 2007 Jul;34(1):94-104. doi: 10.1016/j.jpainsymman.2006.10.015. Epub 2007 May 23. PMID 17509812
- [Background] Stone P, Richards M, Hardy J. Fatigue in patients with cancer. Eur J Cancer. 1998 Oct;34(11):1670-6. doi: 10.1016/s0959-8049(98)00167-1. PMID 9893650
- [Background] Chan CW, Molassiotis A. The impact of fatigue on Chinese cancer patients in Hong Kong. Support Care Cancer. 2001 Jan;9(1):18-24. doi: 10.1007/s005200000192. PMID 11147138
- [Background] Lou Y, Yates P, McCarthy A, Wang H. Fatigue self-management: a survey of Chinese cancer patients undergoing chemotherapy. J Clin Nurs. 2013 Apr;22(7-8):1053-65. doi: 10.1111/jocn.12174. PMID 23480501
- [Background] Curt GA, Breitbart W, Cella D, Groopman JE, Horning SJ, Itri LM, Johnson DH, Miaskowski C, Scherr SL, Portenoy RK, Vogelzang NJ. Impact of cancer-related fatigue on the lives of patients: new findings from the Fatigue Coalition. Oncologist. 2000;5(5):353-60. doi: 10.1634/theoncologist.5-5-353. PMID 11040270
- [Background] Gupta D, Lis CG, Grutsch JF. The relationship between cancer-related fatigue and patient satisfaction with quality of life in cancer. J Pain Symptom Manage. 2007 Jul;34(1):40-7. doi: 10.1016/j.jpainsymman.2006.10.012. Epub 2007 May 25. PMID 17532179
- [Background] Dean A. The holistic management of fatigue within palliative care. Int J Palliat Nurs. 2019 Aug 2;25(8):368-376. doi: 10.12968/ijpn.2019.25.8.368. PMID 31437105
- [Background] Mucke M; Mochamat; Cuhls H, Peuckmann-Post V, Minton O, Stone P, Radbruch L. Pharmacological treatments for fatigue associated with palliative care. Cochrane Database Syst Rev. 2015 May 30;2015(5):CD006788. doi: 10.1002/14651858.CD006788.pub3. PMID 26026155
- [Background] Bower JE. Cancer-related fatigue--mechanisms, risk factors, and treatments. Nat Rev Clin Oncol. 2014 Oct;11(10):597-609. doi: 10.1038/nrclinonc.2014.127. Epub 2014 Aug 12. PMID 25113839
- [Background] Lower EE, Fleishman S, Cooper A, Zeldis J, Faleck H, Yu Z, Manning D. Efficacy of dexmethylphenidate for the treatment of fatigue after cancer chemotherapy: a randomized clinical trial. J Pain Symptom Manage. 2009 Nov;38(5):650-62. doi: 10.1016/j.jpainsymman.2009.03.011. PMID 19896571
- [Background] Bruera E, Yennurajalingam S, Palmer JL, Perez-Cruz PE, Frisbee-Hume S, Allo JA, Williams JL, Cohen MZ. Methylphenidate and/or a nursing telephone intervention for fatigue in patients with advanced cancer: a randomized, placebo-controlled, phase II trial. J Clin Oncol. 2013 Jul 1;31(19):2421-7. doi: 10.1200/JCO.2012.45.3696. Epub 2013 May 20. PMID 23690414
- [Background] Golden RN, Gaynes BN, Ekstrom RD, Hamer RM, Jacobsen FM, Suppes T, Wisner KL, Nemeroff CB. The efficacy of light therapy in the treatment of mood disorders: a review and meta-analysis of the evidence. Am J Psychiatry. 2005 Apr;162(4):656-62. doi: 10.1176/appi.ajp.162.4.656. PMID 15800134
- [Background] NCCN Guidelines Version 2.2018 Cancer-Related Fatigue, page 26/64. 2018.
- [Background] Thong MSY, van Noorden CJF, Steindorf K, Arndt V. Cancer-Related Fatigue: Causes and Current Treatment Options. Curr Treat Options Oncol. 2020 Feb 5;21(2):17. doi: 10.1007/s11864-020-0707-5. PMID 32025928
- [Background] Phipps-Nelson J, Redman JR, Dijk DJ, Rajaratnam SM. Daytime exposure to bright light, as compared to dim light, decreases sleepiness and improves psychomotor vigilance performance. Sleep. 2003 Sep;26(6):695-700. doi: 10.1093/sleep/26.6.695. PMID 14572122
- [Background] Lam RW, Levitt AJ, Levitan RD, Michalak EE, Cheung AH, Morehouse R, Ramasubbu R, Yatham LN, Tam EM. Efficacy of Bright Light Treatment, Fluoxetine, and the Combination in Patients With Nonseasonal Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Jan;73(1):56-63. doi: 10.1001/jamapsychiatry.2015.2235. PMID 26580307
- [Background] Sit DK, McGowan J, Wiltrout C, Diler RS, Dills JJ, Luther J, Yang A, Ciolino JD, Seltman H, Wisniewski SR, Terman M, Wisner KL. Adjunctive Bright Light Therapy for Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2018 Feb 1;175(2):131-139. doi: 10.1176/appi.ajp.2017.16101200. Epub 2017 Oct 3. PMID 28969438
- [Background] Bernatchez MS, Savard J, Ivers H. Disruptions in sleep-wake cycles in community-dwelling cancer patients receiving palliative care and their correlates. Chronobiol Int. 2018 Jan;35(1):49-62. doi: 10.1080/07420528.2017.1381615. Epub 2017 Nov 16. PMID 29144172
- [Background] Liu L, Marler MR, Parker BA, Jones V, Johnson S, Cohen-Zion M, Fiorentino L, Sadler GR, Ancoli-Israel S. The relationship between fatigue and light exposure during chemotherapy. Support Care Cancer. 2005 Dec;13(12):1010-7. doi: 10.1007/s00520-005-0824-5. Epub 2005 Apr 29. PMID 15864659
- [Background] Jeste N, Liu L, Rissling M, Trofimenko V, Natarajan L, Parker BA, Ancoli-Israel S. Prevention of quality-of-life deterioration with light therapy is associated with changes in fatigue in women with breast cancer undergoing chemotherapy. Qual Life Res. 2013 Aug;22(6):1239-44. doi: 10.1007/s11136-012-0243-2. Epub 2012 Aug 3. PMID 22865153
- [Background] Ancoli-Israel S, Rissling M, Neikrug A, Trofimenko V, Natarajan L, Parker BA, Lawton S, Desan P, Liu L. Light treatment prevents fatigue in women undergoing chemotherapy for breast cancer. Support Care Cancer. 2012 Jun;20(6):1211-9. doi: 10.1007/s00520-011-1203-z. Epub 2011 Jun 11. PMID 21660669
- [Background] Redd WH, Valdimarsdottir H, Wu LM, Winkel G, Byrne EE, Beltre MA, Liebman ES, Erazo T, Hayes JA, Isola L, Scigliano E, Meschian Y, Lutgendorf S, Ancoli-Israel S. Systematic light exposure in the treatment of cancer-related fatigue: a preliminary study. Psychooncology. 2014 Dec;23(12):1431-4. doi: 10.1002/pon.3553. Epub 2014 May 2. No abstract available. PMID 24798589
- [Background] Johnson JA, Garland SN, Carlson LE, Savard J, Simpson JS, Ancoli-Israel S, Campbell TS. The LITE study: Rationale and protocol for a randomized controlled trial of light therapy for cancer-related fatigue in cancer survivors. Contemp Clin Trials. 2016 Jul;49:166-73. doi: 10.1016/j.cct.2016.07.004. Epub 2016 Jul 6. PMID 27394380
- [Background] Johnson JA, Garland SN, Carlson LE, Savard J, Simpson JSA, Ancoli-Israel S, Campbell TS. Bright light therapy improves cancer-related fatigue in cancer survivors: a randomized controlled trial. J Cancer Surviv. 2018 Apr;12(2):206-215. doi: 10.1007/s11764-017-0659-3. Epub 2017 Nov 10. PMID 29127575
- [Background] Stockler MR, O'Connell R, Nowak AK, Goldstein D, Turner J, Wilcken NR, Wyld D, Abdi EA, Glasgow A, Beale PJ, Jefford M, Dhillon H, Heritier S, Carter C, Hickie IB, Simes RJ; Zoloft's Effects on Symptoms and survival Time Trial Group. Effect of sertraline on symptoms and survival in patients with advanced cancer, but without major depression: a placebo-controlled double-blind randomised trial. Lancet Oncol. 2007 Jul;8(7):603-12. doi: 10.1016/S1470-2045(07)70148-1. PMID 17548243
- [Background] Dev R D-GM, De La Cruz M, Rhondali W, Hui D, Bruer E. Feasibility of a Randomized Controlled Trial of Light Therapy in Cancer Patients with Insomnia. Journal of Palliative Care & Medicine. 2014;04(04).
- [Background] Chen EK, Riffin C, Reid MC, Adelman R, Warmington M, Mehta SS, Pillemer K. Why is high-quality research on palliative care so hard to do? Barriers to improved research from a survey of palliative care researchers. J Palliat Med. 2014 Jul;17(7):782-7. doi: 10.1089/jpm.2013.0589. Epub 2014 Jun 2. PMID 24885960
- [Background] Higginson IJ. Research challenges in palliative and end of life care. BMJ Support Palliat Care. 2016 Mar;6(1):2-4. doi: 10.1136/bmjspcare-2015-001091. No abstract available. PMID 26893386
- [Background] Higginson IJ, Evans CJ, Grande G, Preston N, Morgan M, McCrone P, Lewis P, Fayers P, Harding R, Hotopf M, Murray SA, Benalia H, Gysels M, Farquhar M, Todd C; MORECare. Evaluating complex interventions in end of life care: the MORECare statement on good practice generated by a synthesis of transparent expert consultations and systematic reviews. BMC Med. 2013 Apr 24;11:111. doi: 10.1186/1741-7015-11-111. PMID 23618406